CLINICAL TRIAL: NCT07268365
Title: Is Cap Assisted Endoscopy Useful in Acute Upper Gastrointestinal Bleeding ?
Acronym: CAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2025_843_0158
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Cap-assisted Endoscopy; Upper Gastro Intestinal Bleeding; Endoscopy
Keywords: Cap-assisted endoscopy; upper gastro intestinal bleeding; endoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard upper endoscopy (Active Comparator): standard upper endoscopy
  Interventions: Procedure: upper endoscopy
- CAP (Experimental): upper endoscopy with the placement of an endoscopic cap
  Interventions: Procedure: upper endoscopy; Procedure: CAP

INTERVENTIONS:
Procedure: upper endoscopy — All patients with the inclusion criteria will be randomized (randomization 1:1) to undergo either an upper endoscopy with an endoscopic cap or without a cap
Procedure: CAP — All patients with the inclusion criteria will be randomized (randomization 1:1) to undergo either an upper endoscopy with an endoscopic cap or without a cap
  Arms: CAP

SUMMARY:
High digestive bleeding (HDH) is a medical emergency associated with high morbidity and mortality rates and significant healthcare costs. Upper endoscopy can locate the bleeding and treat it. However, the source of bleeding can be difficult to identify, even for the most experienced endoscopists, due to the location of the bleeding (posterior wall of the bulb, gastric or duodenal folds, papillary region, esophagogastric junction), instability of the tube due to gastric and pyloric contractions and respiratory movements, leading to longer procedure times, hemostasis failure, or even the absence of bleeding visualization. The use of a cap attached to the endoscope facilitates exploration of blind areas of the colonic mucosa located behind folds, thus reducing the rate of missed polyps and cecal intubation time. To date, there is no study evaluating the systematic use of a cap in patients with suspected high digestive bleeding. A series of four cases demonstrated its benefit, allowing for better exposure of the bleeding lesion, better unfolding of intestinal folds, and thus a more effective and quicker hemostatic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Upper GI bleeding suspected in presence of melena or hematemesis
* Glasgow Blatchford score > 8
* Upper gastroscopy at Amiens University Hospital
* Follow-up at Amiens university hospital
* Presence of gastric or duodenal ulcer requiring endoscopic hemostasis (FORREST Ia, Ib, IIa, IIb)
* No opposition to the study
* No guardianship or curators

Exclusion Criteria:

* Patient with clinical suspicion of portal hypertension
* Known liver failure
* Patient with digestive hemorrhage related to a lesion located beyond the 2nd duodenum
* Patient with digestive hemorrhage related to a varicose lesion (esophageal or gastric varices)
* Patient with bleeding associated with esophagitis
* Patient with bleeding associated with angiodysplasias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
procedure time until endoscopic hemostasis is achieved | 1 month
  procedure time until endoscopic hemostasis is achieved

SECONDARY OUTCOMES:
therapeutic success rate | 1 month
  therapeutic success rate
clinical success rate | 1 month
  clinical success rate
time until bleeding localization | up to 1 month
  time until bleeding localization
duration of hemostasis achievement | up to 1 month
  duration of hemostasis achievement
endoscope stability | up to 1 month
  assessment of endoscopist satisfaction in terms of endoscope stability
lesion visualization | up to 1 month
  lesion visualization
hemostasis | up to 1 month
  hemostasis

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No